CLINICAL TRIAL: NCT05759351
Title: Appendectomy During Pregnancy in General Anesthesia With Perioperative Management Does Not Influence Normal Child Development: 10-year Study
Brief Title: Appendectomy During Pregnancy and Child Development
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Branko Bogdanic, MD, PhD, Clinical Hospital Centre Zagreb
Other Study IDs: 202201
Record Dates: First submitted 2023-01-01; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Appendicitis Acute; Pregnancy Related; Anesthetic Toxicity; Child Development; Psychomotor Development Impaired
Keywords: appendicitis, pregnancy, child development, psychomotor development impaired
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Maternal acute appendicitis during pregnancy is the most common abdominal surgical emergency. Long-term neurodevelopmental issues were scarcely reported. The aim of the study is to investigate the impact of appendicitis and appendectomy during pregnancy in general anesthesia on the cognitive and psychomotor development of children.

DETAILED DESCRIPTION:
Maternal acute appendicitis (AA) is the most common emergent abdominal surgical condition during pregnancy. Brain development in a fetus is dynamic and complex, and therefore much more vulnerable to different agents. Gastrointestinal operations during pregnancy are performed in general anesthesia and anesthetic neurotoxicity in the developing brain, through the period from a fetus to a child, delivered inconsistent results.

Child development after AA or other intra-abdominal inflammatory/infective condition during pregnancy was not consistently reported or studied. In most reports, the length of fetal follow-up after appendectomy for AA during pregnancy is not defined, not stated, or declared as 'uneventful'.

Investigators will make a study with a structured children's cognitive and neurodevelopmental follow-up whose mothers had operated acute appendicitis during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women operated for acute appendicitis (January 2006- December 2020)

Exclusion Criteria:

* pregnant women younger than 18
* nonpregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant women operated for acute appendicitis at the University Hospital Center Zagreb, Croatia, January 2006- December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Impact of maternal sociodemographic characteristics and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include maternal sociodemographic characteristics- chronic diseases, psychiatric diseases, childhood disease, level of education, level of partner's education, working status, marital status, city or rural living, GPA (gravida, para, abortus) status, number of household persons
Impact of obstetric factors and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include obstetric factors- age at delivery, gestational week of delivery, delivery route, elective or emergent delivery, tocolysis, neonatal height, neonatal weight, APGAR score, complications during pregnancy, infections or pyrexias, congenital malformations)
Impact of clinical-laboratory parameters and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include clinical-laboratory parameters- differential blood count, C-reactive protein, platelets, axillary temperature, transabdominal ultrasound, Alvarado score, Tzanakis score)
Impact of surgical factors and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include surgical factors- open or laparoscopic appendectomy, type, and duration of antibiotic therapy, degree of appendiceal inflammation
Impact of anesthesiologic factors and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include anesthesiologic parameters- type and duration of anesthesia, anesthetics and analgesics used, maternal behavior and emotional status during pregnancy (presence and extent of stressful events, alcohol, medication, and/or drugs consumption, smoking, maternal nutrition and diet)
Impact of pediatric factors and inflammation of the appendix and appendectomy during pregnancy under general anesthesia on the cognitive and psychomotor development of children | January 2006 to December 2020
  Analyzed data will include pediatric parameters (child's growth and development, existence of congenital malformations, childhood diseases, medical conditions and procedures, need for surgical treatments, routine pediatric checkups, physical or speech therapy, referrals to specialists, early separations, exposure to highly stressful or traumatic events, and academic success for older children)
  A psychiatry resident will led the interviews using a structured questionnaire for mothers designed for this study during interviews. Based on the parents' observations and assessment and available medical data, the child's psychomotor and cognitive development and medical status will be analyzed during a clinical interview with the mother.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Zagreb, Zagreb, Croatia

REFERENCES:
- [Background] Yang J, Wen SW, Krewski D, Corsi DJ, Walker M, Mattison D, Moog R, McNair D, Huang H, Zhuang G. Association of treatments for acute appendicitis with pregnancy outcomes in the United States from 2000 to 2016: Results from a multi-level analysis. PLoS One. 2021 Dec 13;16(12):e0260991. doi: 10.1371/journal.pone.0260991. eCollection 2021. PMID 34898628
- [Background] Yu CH, Weng SF, Ho CH, Chen YC, Chen JY, Chang YJ, Wang JJ, Wu MP, Chu CC. Pregnancy outcomes following nonobstetric surgery during gestation: a nationwide population-based case-control study in Taiwan. BMC Pregnancy Childbirth. 2018 Nov 26;18(1):460. doi: 10.1186/s12884-018-2079-4. PMID 30477448
- [Background] Choi JJ, Mustafa R, Lynn ET, Divino CM. Appendectomy during pregnancy: follow-up of progeny. J Am Coll Surg. 2011 Nov;213(5):627-32. doi: 10.1016/j.jamcollsurg.2011.07.016. Epub 2011 Aug 19. PMID 21856183
- [Background] Kocael PC, Simsek O, Saribeyoglu K, Pekmezci S, Goksoy E. Laparoscopic surgery in pregnant patients with acute abdomen. Ann Ital Chir. 2015 Mar-Apr;86(2):137-42. PMID 25952362
- [Background] Hannan MJ, Hoque MM, Begum LN. Laparoscopic appendectomy in pregnant women: experience in Chittagong, Bangladesh. World J Surg. 2012 Apr;36(4):767-70. doi: 10.1007/s00268-012-1445-z. PMID 22311138
- [Background] Rizzo AG. Laparoscopic surgery in pregnancy: long-term follow-up. J Laparoendosc Adv Surg Tech A. 2003 Feb;13(1):11-5. doi: 10.1089/109264203321235403. PMID 12676015
- [Background] Al-Haddad BJS, Jacobsson B, Chabra S, Modzelewska D, Olson EM, Bernier R, Enquobahrie DA, Hagberg H, Ostling S, Rajagopal L, Adams Waldorf KM, Sengpiel V. Long-term Risk of Neuropsychiatric Disease After Exposure to Infection In Utero. JAMA Psychiatry. 2019 Jun 1;76(6):594-602. doi: 10.1001/jamapsychiatry.2019.0029. PMID 30840048
- [Background] de Jonge L, Bos HJ, van Langen IM, de Jong-van den Berg LT, Bakker MK. Antibiotics prescribed before, during and after pregnancy in the Netherlands: a drug utilization study. Pharmacoepidemiol Drug Saf. 2014 Jan;23(1):60-8. doi: 10.1002/pds.3492. Epub 2013 Aug 3. PMID 23913654
- [Background] Sumilo D, Nirantharakumar K, Willis BH, Rudge GM, Martin J, Gokhale K, Thayakaran R, Adderley NJ, Chandan JS, Okoth K, Harris IM, Hewston R, Skrybant M, Deeks JJ, Brocklehurst P. Long term impact of prophylactic antibiotic use before incision versus after cord clamping on children born by caesarean section: longitudinal study of UK electronic health records. BMJ. 2022 May 17;377:e069704. doi: 10.1136/bmj-2021-069704. PMID 35580876
- [Background] Lapin B, Piorkowski J, Ownby D, Freels S, Chavez N, Hernandez E, Wagner-Cassanova C, Pelzel D, Vergara C, Persky V. Relationship between prenatal antibiotic use and asthma in at-risk children. Ann Allergy Asthma Immunol. 2015 Mar;114(3):203-7. doi: 10.1016/j.anai.2014.11.014. Epub 2014 Dec 19. PMID 25532738
- [Background] Tomar N, Uldbjerg CS, Bech BH, Burgner DP, Pedersen LH, Miller JE. Prenatal antibiotic exposure and birth weight. Pediatr Obes. 2022 Feb;17(2):e12831. doi: 10.1111/ijpo.12831. Epub 2021 Jun 30. PMID 34192823
- [Background] Cho HW, Cho GJ, Noh E, Hong JH, Kim M, Lee JK. Pregnancy Outcomes Following Laparoscopic and Open Surgery in Pelvis during Pregnancy: a Nationwide Population-based Study in Korea. J Korean Med Sci. 2021 Jul 26;36(29):e192. doi: 10.3346/jkms.2021.36.e192. PMID 34313034
- [Background] Shigemi D, Aso S, Matsui H, Fushimi K, Yasunaga H. Safety of Laparoscopic Surgery for Benign Diseases during Pregnancy: A Nationwide Retrospective Cohort Study. J Minim Invasive Gynecol. 2019 Mar-Apr;26(3):501-506. doi: 10.1016/j.jmig.2018.06.008. Epub 2018 Aug 2. PMID 29909089
- [Background] Bleeser T, Van Der Veeken L, Devroe S, Vergote S, Emam D, van der Merwe J, Ghijsens E, Joyeux L, Basurto D, Van de Velde M, Deprest J, Rex S. Effects of Maternal Abdominal Surgery on Fetal Brain Development in the Rabbit Model. Fetal Diagn Ther. 2021;48(3):189-200. doi: 10.1159/000512489. Epub 2021 Feb 25. PMID 33631746
- [Background] Augustin G, Boric M, Barcot O, Puljak L. Discordant outcomes of laparoscopic versus open appendectomy for suspected appendicitis during pregnancy in published meta-analyses: an overview of systematic reviews. Surg Endosc. 2020 Oct;34(10):4245-4256. doi: 10.1007/s00464-020-07674-6. Epub 2020 Jun 16. PMID 32556754
- [Background] Tekin A, Evruke C, Deveci O. Maternal and fetal near-term sheep cytokine responses to carbon dioxide pneumoperitoneum. Surg Laparosc Endosc Percutan Tech. 2009 Apr;19(2):138-41. doi: 10.1097/SLE.0b013e31819756bf. PMID 19390281
- [Background] de la Fuente SG, Pinheiro J, Gupta M, Eubanks WS, Reynolds JD. Early postnatal behavior deficits after maternal carbon dioxide pneumoperitoneum during pregnancy. Surg Endosc. 2003 Nov;17(11):1823-5. doi: 10.1007/s00464-002-8871-1. Epub 2003 Jun 17. PMID 12802645
- [Background] Andropoulos DB. Effect of Anesthesia on the Developing Brain: Infant and Fetus. Fetal Diagn Ther. 2018;43(1):1-11. doi: 10.1159/000475928. Epub 2017 Jun 7. PMID 28586779
- [Background] Bleeser T, Van Der Veeken L, Fieuws S, Devroe S, Van de Velde M, Deprest J, Rex S. Effects of general anaesthesia during pregnancy on neurocognitive development of the fetus: a systematic review and meta-analysis. Br J Anaesth. 2021 Jun;126(6):1128-1140. doi: 10.1016/j.bja.2021.02.026. Epub 2021 Apr 6. PMID 33836853
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Walkden GJ, Gill H, Davies NM, Peters AE, Wright I, Pickering AE. Early Childhood General Anesthesia and Neurodevelopmental Outcomes in the Avon Longitudinal Study of Parents and Children Birth Cohort. Anesthesiology. 2020 Nov 1;133(5):1007-1020. doi: 10.1097/ALN.0000000000003522. PMID 32898216